CLINICAL TRIAL: NCT04333706
Title: A Dose Finding Phase 1 of Sarilumab Plus Capecitabine in HER2/Neu-Negative Metastatic Breast Cancer and a Single-arm, Historically-controlled Phase 2 Study of Sarilumab Plus Capecitabine in Stage I-III Triple Negative Breast Cancer With High-Risk Residual Disease (EMPOWER)
Acronym: EMPOWER
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Southern California (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1B-22-3; HS-23-00019 (Other: USC IRB); 1R01CA238387-01A1 (NIH)
Record Dates: First submitted 2020-04-01; First posted 2020-04-03 (Actual); Last update posted 2025-04-17 (Actual); Status verified 2025-04

CONDITIONS: Breast; Metastatic; Triple Negative; Cancer; Disseminated Tumor Cell
MeSH Terms: conditions — Neoplasm Metastasis; Neoplasms | interventions — Capecitabine; sarilumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Experimental: Phase I (Experimental): A dose finding study of sarilumab plus capecitabine in patients with metastatic TNBC and metastatic HER2/neu-negative and hormone resistant breast cancer.
  Interventions: Combination Product: Sarilumab 150mg or 200 mg plus Capecitabine; Combination Product: Sarilumab 150mg plus Capecitabine
- Phase 2 single arm study (Experimental): Study of adjuvant sarilumab plus capecitabine in stage I to III TNBC with less than a pCR
  Interventions: Combination Product: Sarilumab 150mg or 200 mg plus Capecitabine; Combination Product: Sarilumab 150mg plus Capecitabine
- Parallel Baseline Arm (Other): Study of standard adjuvant capecitabine in stage I to III TNBC with less than a pCR. This Arm will be open in parallel with both Phases 1 and 2. Blood samples will be obtained during the course of the study. Bone marrow samples are optional.
  Interventions: Drug: Capecitabine

INTERVENTIONS:
Drug: Capecitabine — Capecitabine 1000 mg BID
  Arms: Parallel Baseline Arm
Combination Product: Sarilumab 150mg or 200 mg plus Capecitabine — Sarilumab 150mg or 200 mg plus Capecitabine 1000 mg BID
  Arms: Experimental: Phase I; Phase 2 single arm study
Combination Product: Sarilumab 150mg plus Capecitabine — Dose escalation schedule of sarilumab. The starting dose for sarilumab is 150 mg SQ every 21 days, given 3 days prior to the first 4 of 8 cycles of capecitabine 1000 mg BID.
  Arms: Experimental: Phase I; Phase 2 single arm study

SUMMARY:
This study looks to advance a novel and potent strategy to eliminate minimal residual disease (MRD) in triple negative breast cancer (TNBC) present even after multimodal treatment, thereby improving survival and increasing cure rate in this aggressive cancer. Patients with locally advanced TNBC are at high risk of developing lethal metastatic disease within 2 years of diagnosis, especially for those without a pathologic complete response (pCR) after neoadjuvant chemotherapy. The high risk occurs despite surgical excision of the primary tumor and axillary lymph nodes to eliminate residual disease.

DETAILED DESCRIPTION:
The study will consist of two phases, I and II.

Phase I will include patients with metastatic TNBC, HER2/neu-negative and hormone resistant breast cancer. A total of 4 doses of sarilumab will be given with the starting dose of 150 mg SQ at 3-weeks cycles given 3 days prior to each of the first 4 of 8 cycles of capecitabine (1000 mg/m2/BID; for 14 days every 21 days). If dose escalation is possible, sarilumab will be administered every 3 weeks at 200 mg SQ for 4 doses. Blood samples will be obtained prior during the course of treatment. Bone marrow samples are optional.

Phase II is a single arm study in Stage I to III TNBC with less than a complete pCR after neoadjuvant therapy evaluating the combination of sarilumab with capecitabine (1000mg/m2/BID; for 14 days every 21 days) as compared to historical control patients treated with capecitabine alone. There are 8 cycles of capecitabine. The first 4 cycles will be combined with sarilumab. The Phase II sarilumab dose will be determined by the Phase I best tolerated dose. Blood samples will be obtained prior during the course of treatment. Bone marrow samples are optional.

A pilot parallel biological baseline study of standard adjuvant capecitabine in stage I to III TNBC with less than a pCR will be performed. This Arm will be open in parallel with both Phases 1 and 2. Blood samples will be obtained prior during the course of treatment. Bone marrow samples are optional.

ELIGIBILITY:
Inclusion Criteria:

* A. Written informed consent obtained from the subject and the ability for the subject to comply with all the study-related procedures.
* B. Both males and females ≥ eighteen years of age
* C. A clinical diagnosis of metastatic triple negative or hormone resistant, Her2/neu-negative breast cancer that has been confirmed histologically at one point during the course of the disease. TNBC is defined as ER/PR IHC positivity rate of <10% and Her2Neu-negative (Phase I only)
* D. A life expectancy of at least 6 months. (Phase I only)
* E. Any previous cytotoxic chemotherapy must have been a minimum of 3 weeks prior to study drug administration. There is no limit on the number of prior therapies. For ER/PR-positive tumors, endocrine therapy must have been included in at least one of those prior regimens. Prior capecitabine is allowed only if not given in the treatment regimen immediately prior to the enrollment in this study. (Phase I only)
* F. A diagnosis of TNBC confirmed histologically and defined as ER/PR IHC positivity rate of <10% and Her2/neu-negative. (Phase II and Parallel Baseline Arm only)
* G. A pathologic confirmation of stage I, or II, or III breast cancer with less than a complete pCR, defined as the absence of residual invasive cancer in resected breast specimen and sampled lymph nodes with residual noninvasive cancer or in situ disease allowed. (Phase II and Parallel Baseline Arm only)
* H. Must not have received prior systemic treatment for breast cancer except for those included in the neoadjuvant regimen and the neoadjuvant regimen must not have included capecitabine nor sarilumab. (Phase II and Parallel Baseline Arm only)
* I. An ECOG Performance Status ≤2.
* J. Adequate organ function defined as:

  1. Absolute neutrophil count (ANC) > 1500/mcl (use of G-CSF is allowed)
  2. Platelets ≥ 100,000/mcl
  3. Hemoglobin ≥ 9 (pRBC +/- ESA are allowed)
  4. ALT ≤ 5 x ULN
  5. AST ≤ 5 x ULN
  6. Bilirubin ≤ 3 x ULN
  7. GFR ≥ 30 ml/min
* K. Women of childbearing potential (WOCBP) must be using a highly effective method of contraception to avoid pregnancy throughout the study and for at least 24 weeks after the last dose of study drug to minimize the risk of pregnancy. Prior to study enrollment, women of childbearing potential must be advised of the importance of avoiding pregnancy during trial participation and the potential risk factors for an unintentional pregnancy.
* L. Males with female partners of child-bearing potential must agree to use physician-approved contraceptive methods (e.g., abstinence, condoms, vasectomy) throughout the study and should avoid conceiving children for 24 weeks following the last dose of study drug.

Exclusion Criteria:

* A. Females or males of childbearing potential who are unwilling or unable to use an acceptable method to avoid pregnancy for the entire study period and for at least 24 weeks after the last dose of study drug.
* B. Females who are pregnant or breastfeeding.
* C. History of any other disease, metabolic dysfunction, physical examination finding, or clinical laboratory finding giving reasonable suspicion of a disease or condition that contraindicates the use of protocol therapy or that might affect the interpretation of the results of the study or that puts the subject at high risk for treatment complications, in the opinion of the treating physician.
* D. Hepatitis B infection except for prior vaccination. (Phase I and Phase II only).
* E. Known history of tuberculosis injection. (Phase I and Phase II only).
* F. A history of diverticulitis. (Phase I and Phase II only).
* G. Use of live vaccines within 30 days prior to study treatment due to the risk of infection. Examples of live vaccines include, but are not limited to, the following: measles, mumps, rubella (MMR), varicella/zoster (chicken pox), yellow fever, rabies, Bacillus Calmette-Guérin (BCG), and typhoid vaccine. Seasonal influenza vaccines for injection are generally killed virus vaccines and are allowed; however, intranasal influenza vaccines (e.g. FluMist) are live attenuated vaccines and are not allowed. (Phase I and Phase II only)
* H. History of other malignancy that in the primary oncologist's estimation has at the time of study participation a higher risk of recurrence or death than the study-related cancer.
* I. Prisoners or subjects who are involuntarily incarcerated.
* J. Subjects who are compulsorily detained for treatment of either a psychiatric or physical illness.
* K. Subjects demonstrating an inability to comply with the study and/or follow-up procedures.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Estimated)
Dates: Start 2020-09-26 (Actual); Primary Completion 2026-09-01 (Estimated); Study Completion 2027-09-01 (Estimated)

PRIMARY OUTCOMES:
Phase I: Maximum Tolerated Dose (MTD) | first treatment up to 9 weeks
  Establish MTD of sarilumab plus capecitabine in patients with metastatic TNBC and metastatic HER2/neu-negative and hormone resistant breast cancer
Phase I: Dose-limiting toxicity (DLT) | first treatment up to 9 weeks
  Defined events that are possibly, probably, or definitely related to the study treatment:
Phase II:To determine the percent of patients with positive CTCs and DTCs (if available) becoming negative CTCs and DTCs (if available) after treatment | baseline up to 14 weeks
  Bone marrow aspirates will be performed before treatment and at defined time points during treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Priya Jayachandran, MD, Principal Investigator — University of Southern California
Locations (3):
- United States (3):
  - Los Angeles General Medical Center, Los Angeles, California
  - USC/Norris Comprehensive Cancer Center, Los Angeles, California
  - UF Health, Gainesville, Florida

IPD SHARING:
Plan to Share IPD: No